CLINICAL TRIAL: NCT06074016
Title: Pharmacokinetic Model Based on Population Physiology of Oral and Intranasal Formulations of Zolmitriptan in Healthy Volunteers
Brief Title: Pharmacokinetics in Oral and Intranasal Formulations of Zolmitriptan.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IMIMFCTL/ZOL_1
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — zolmitriptan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zolmitriptan intranasal. (Experimental)
  Interventions: Drug: Zolmitriptan intranasal.
- Zolmitriptan oral. (Experimental)
  Interventions: Drug: Zolmitriptan oral.

INTERVENTIONS:
Drug: Zolmitriptan intranasal. — Zolmitriptan nasal spray is supplied in a single-use, ready-to-use spray unit. It is administered in one nostril. The full protocol will explain how to use it. Following drug administration, study subjects will continue to fast for a minimum of 4h and snacks and standard meals may be served at scheduled times after drug administration (snack: +4h; lunch: +7h; snack: +10h). Liquid intake will not be allowed from 2h before to 2h after drug administration.
  Arms: Zolmitriptan intranasal.
Drug: Zolmitriptan oral. — Zolmitriptan 5 mg orally disintegrating tablet is to be taken without liquids. For oral administration, each tablet will be placed in the top of the tongue without any liquid and will disperse in a matter of seconds, then be swallowed with saliva. Following drug administration, study subjects will continue to fast for a minimum of 4h and snacks and standard meals may be served at scheduled times after drug administration (snack: +4h; lunch: +7h; snack: +10h). Liquid intake will not be allowed from 2h before to 2h after drug administration.
  Arms: Zolmitriptan oral.

SUMMARY:
This is a phase I study to evaluate the PBPK of zolmitriptan intranasal versus oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers by physical examination, vital signs, ECG, and safety laboratory parameters and results must be within normal ranges or considered not clinically relevant by the investigator.
* Age ≥ 18 years and ≤ 55 years.
* Body mass index (BMI) ≥ 18 and ≤ 30.
* Able/willing to accept restrictions regarding diet, physical exercise, and consumption of alcohol and/or xanthine-containing items when outside the Clinical Research Unit (CRU)
* Able to read Spanish and adhere to study requirements.
* Informed consent signed before any procedure required by the study.

Exclusion Criteria:

* Smoking.
* History or clinically relevant diseases.
* Be under administrative or legal supervision.
* Pregnancy and breastfeeding.
* Positive blood or urine drug of abuse test or breathalyzer prior to study drug administration.
* Any history, disease, disorder, condition, anomaly or clinical finding that is relevant in the judgment of the investigator that may interfere with the study.
* Known hypersensitivity to any drug or excipient of the drug.
* Use of medications, inhibitors, any prescription or over-the-counter products, including herbs, homeopathy, vitamins, minerals, and nutritional supplements, before or during the study, that may interfere with the conduct and results of the study.
* Donation or transfusion of blood or plasma before, during or after study drug administration.
* History of inadequate venous access and/or experience of difficulty donating blood.
* Not being able/unwilling to accept restrictions regarding diet, physical exercise and consumption of alcohol and/or articles containing xanthine when outside the CRU.
* Subject included in a clinical study in the 3 months prior to the study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Effects of zolmitriptan on heart rate (HR). | Up to 24 hours.
Effects of zolmitriptan on systolic and diastolic blood pressure (BP). | Up to 24 hours.

SECONDARY OUTCOMES:
Concentration of zolmitriptan on vasoactive intestinal polypeptide (VIP) in captures Day 1. | Up to 24 hours.

OTHER OUTCOMES:
Adverse effects. | Up to 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain